CLINICAL TRIAL: NCT00054587
Title: Randomized And Multicentric Opened Phase III Study Evaluating The Concomitant Administration Of Docetaxel 75MG/M2 and Epirubicine 75MG/M2 Versus FEC 100 In Non Metastatic With Positive Lymphatic Nodes Breast Cancer Subjects, And The Sequential Addition Of Herceptin In (HER2+++) And (HER2++ And FISH+) Subjects
Brief Title: Combination Chemotherapy With or Without Trastuzumab in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0140/0005 - PACS 04; FRE-FNCLCC-PACS-04/0005; EU-20236; PACS04 (Other: UNICANCER)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 FEC (Active Comparator): Patients receive fluorouracil IV, or epirubicin IV, and cyclophosphamide IV on day 1. Treatment repeats every 3 weeks for 6 courses. Patients then undergo radiotherapy 5 days a week for 5 weeks.
  Interventions: Biological: Trastuzumab; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Fluorouracil
- 6 DE (Experimental): Patients receive epirubicin IV over 10 minutes and docetaxel IV over 1 hour on day 1. Treatment repeats every 3 weeks for 6 courses. Patients then undergo radiotherapy as in arm I
  Interventions: Biological: Trastuzumab; Drug: docetaxel; Drug: Epirubicin

INTERVENTIONS:
Biological: Trastuzumab — 8 mg/kg at month M6, followed by a maintenance dose of 6 mg/kg every 3 weeks for a 1 year (i.e. 18 injections in total)
  Other Names: Herceptin
Drug: Cyclophosphamide — 500 mg/m², D1 and every 3 weeks
  Arms: 6 FEC
Drug: docetaxel — on day D1 of each cycle : dose: 75 mg/m², route: i.v. injection over 1 hour, every 3 weeks
  Arms: 6 DE
Drug: Epirubicin — 100 mg/m², D1 and every 3 weeks
  Other Names: epirubicin hydrochloride
Drug: Fluorouracil — 500 mg/m², D1 and every 3 weeks
  Arms: 6 FEC

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which regimen of chemotherapy plus radiation therapy with or without trastuzumab is more effective in treating breast cancer.

PURPOSE: Randomized phase III trial to compare two different chemotherapy regimens plus radiation therapy with or without trastuzumab in treating women who have breast cancer that has spread to lymph nodes in the axilla (under the arm).

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of adjuvant cyclophosphamide, epirubicin, and fluorouracil vs adjuvant docetaxel and epirubicin, in terms of 5-year survival without relapse, in women with nonmetastatic adenocarcinoma of the breast with lymph node invasion.
* Determine survival of patients treated with these regimens.
* Compare the tolerability of trastuzumab (Herceptin) in patients treated with these regimens.
* Determine the efficacy and tolerability of trastuzumab in patients with hormone receptor-positive tumors.
* Evaluate the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center. Patients are treated in 2 parts.

* Part I: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive fluorouracil IV, or epirubicin IV, and cyclophosphamide IV on day 1. Treatment repeats every 3 weeks for 6 courses. Patients then undergo radiotherapy 5 days a week for 5 weeks.
  * Arm II: Patients receive epirubicin IV over 10 minutes and docetaxel IV over 1 hour on day 1. Treatment repeats every 3 weeks for 6 courses. Patients then undergo radiotherapy as in arm I.

Patients with HER2/neu-positive tumors then proceed to part II. Patients with HER2/neu-negative tumors receive no further treatment.

Patients with hormone (estrogen or progesterone) receptor-positive tumors also receive oral tamoxifen daily beginning after chemotherapy is completed and continuing for 5 years.

* Part II: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive trastuzumab (Herceptin) IV over 30-90 minutes every 3 weeks for 1 year.
  * Arm II: Patients are followed without treatment. Patients not receiving trastuzumab are followed at 4 months, 6 months, every 4 months for 1 year, and then every 6 months for 3 years. Patients receiving trastuzumab are followed at 4 months and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 2,600 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed nonmetastatic, unilateral adenocarcinoma of the breast

  * Axillary lymph node invasion (N1, N2, or N3)
  * No cutaneous invasion
  * No T4a or greater disease
* No clinically or radiologically suspected metastases
* No clinically or radiologically suspected contralateral lesion
* No deeply adherent or inflammatory disease
* Complete surgical resection performed, including removal of at least 5 lymph nodes, and with no residual tumor, within the past 42 days
* No prior breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 to 64

Sex

* Female

Menopausal status

* Not specified

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* ALT and AST no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* Bilirubin no greater than ULN
* Hepatitis B and hepatitis C negative
* No hepatic dysfunction

Renal

* Creatinine less than 1.3 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular

* ECHO normal
* LVEF at least 50%

Pulmonary

* FEV normal
* No dyspnea at rest
* No supplemental oxygen dependence

Other

* Not pregnant
* Fertile patients must use effective contraception
* HIV negative
* No active infection
* No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No contraindication to anthracycline therapy
* No chronic medical or psychological condition
* No geographic or social reason that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy
* No other concurrent chemotherapy
* No contraindication to anthracycline therapy

Endocrine therapy

* No prior hormonal therapy

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 4 weeks since prior experimental therapy

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3010 (Actual)
Dates: Start 2001-06; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 5 years from randomization

SECONDARY OUTCOMES:
Herceptin safety | 5 years from randomization
Overall survival | 5 years from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Marc Spielmann, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (29):
- France (29):
  - Centre Paul Papin, Angers
  - Centre Hospitalier d'Annecy, Annecy
  - Institut Bergonie, Bordeaux
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Intercommunal De Creteil, Créteil
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Institut Prive de Cancerologie, Grenoble
  - Clinique du Petit Colmouilins, Harfleur
  - Centre Hospitalier de Lagny, Lagny-sur-Marne
  - Hopital Andre Mignot, Le Chesnay
  - CMC Les Ormeaux, Le Havre
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Hospitalier Regional Metz Thionville, Metz
  - Centre Hospitalier General Andre Boulloche, Montbéliard
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Hopital Avicenne, Paris
  - Clinique Saint - Pierre, Perpignan
  - CHU Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Clinique Sainte Clotilde, Sainte Clotilde
  - Centre Paul Strauss, Strasbourg
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Mancini J, Genre D, Dalenc F, Maylevin F, Martin AL, Viens P, Julian-Reynier C. Transparency in the presentation of trial results may not increase patients' trust in medical researchers. Clin Trials. 2012 Feb;9(1):90-3. doi: 10.1177/1740774511427063. Epub 2011 Nov 2. PMID 22049088
- [Result] Roché H, Allouache D, Romieu G, et al.: Five-year analysis of the FNCLCC-PACS04 trial: FEC100 vs ED75 for the adjuvant treatment of node positive breast cancer. [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-602, 2009.
- [Result] Spielmann M, Roche H, Delozier T, Canon JL, Romieu G, Bourgeois H, Extra JM, Serin D, Kerbrat P, Machiels JP, Lortholary A, Orfeuvre H, Campone M, Hardy-Bessard AC, Coudert B, Maerevoet M, Piot G, Kramar A, Martin AL, Penault-Llorca F. Trastuzumab for patients with axillary-node-positive breast cancer: results of the FNCLCC-PACS 04 trial. J Clin Oncol. 2009 Dec 20;27(36):6129-34. doi: 10.1200/JCO.2009.23.0946. Epub 2009 Nov 16. PMID 19917839
- [Result] Spielmann M, Roché H, Humblet Y, et al.: 3-year follow-up of trastuzumab following adjuvant chemotherapy in node positive HER2-positive breast cancer patients: results of the PACS-04 trial. [Abstract] Breast Cancer Res Treat 106 (1): A-72, S19, 2007.
- [Result] Spielmann M, Roché H, Delozier T, et al.: Safety analysis from PACS 04--a phase III trial comparing 6 cycles of FEC100 with 6 cycles of ET75 for node-positive early breast cancer patients, followed by sequential trastuzumab in HER2+patients: preliminary results. [Abstract] J Clin Oncol 24 (Suppl 18): A-632, 2006.
- [Derived] O'Sullivan CC, Bradbury I, Campbell C, Spielmann M, Perez EA, Joensuu H, Costantino JP, Delaloge S, Rastogi P, Zardavas D, Ballman KV, Holmes E, de Azambuja E, Piccart-Gebhart M, Zujewski JA, Gelber RD. Efficacy of Adjuvant Trastuzumab for Patients With Human Epidermal Growth Factor Receptor 2-Positive Early Breast Cancer and Tumors </= 2 cm: A Meta-Analysis of the Randomized Trastuzumab Trials. J Clin Oncol. 2015 Aug 20;33(24):2600-8. doi: 10.1200/JCO.2015.60.8620. Epub 2015 Jun 22. PMID 26101239